CLINICAL TRIAL: NCT06342336
Title: Single Arm, Phase I Clinical Study of HS-IT101 Injection in the Treatment of Advanced Solid Tumors
Brief Title: HS-IT101 Injection in the Treatment of Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Qingdao Sino-Cell Biomedicine Co., Ltd. (Industry)
Collaborators: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other); The First Hospital of Jilin University (Other); West China Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HS-IT101ST01-I
Record Dates: First submitted 2024-03-19; First posted 2024-04-02 (Actual); Last update posted 2024-04-02 (Actual); Status verified 2024-03

CONDITIONS: Solid Tumor

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HS-IT101 monotherapy (Experimental): Adoptive transfer of 5x10^9-6x10^10 autologous TIL to patients i.v. in 30-60 minutes.
  Interventions: Drug: HS-IT101 Injection

INTERVENTIONS:
Drug: HS-IT101 Injection — Adoptive transfer of 5x10^9-6x10^10 autologous TIL to patients i.v. in 30-60 minutes.
  Other Names: HS-IT101

SUMMARY:
Single-arm, open-label,interventional study evaluating adoptive cell therapy (ACT) with autologous tumor-infiltrating lymphocyte (TIL) infusion (HS-IT101) after lymphodepletion preparative with fludarabine and cyclophosphamide regimen, followed by IL-2, for the treatment of patients with advanced solid tumor.

DETAILED DESCRIPTION:
HS-IT101 is an adoptive cell transfer therapy that utilizes an autologous TIL manufacturing process, for the treatment of patients with advanced solid tumor. The cell transfer therapy used in this study involves patients receiving lymphodepletion treatment with fludarabine and cyclophosphamide, followed by infusion of autologous TIL, then finnaly followed by the administration of a regimen of IL-2.

ELIGIBILITY:
Inclusion Criteria:

* To be eligible for the study, patients must meet ALL of the following criteria prior to participation:

  1. Age: 18 years to 75 years at the time of consent;
  2. Histologically or cytological diagnosed as advanced soild tumor:
  3. At least one resectable lesion that has not received radiotherapy or other local therapy within 28 days, and the weight of the tissue must be ≥ 0.050g；or resectable lesions capable of producing sufficient TIL;
  4. At least one measurable target lesion, as defined by RECIST v1.1，that has not received radiotherapy or other local therapy unless these therapies occurred 28 days ago and target lesion shows significant progression;
  5. ECOG score 0-1;
  6. Expected life-span more than 3 months;
  7. Adequate organ and bone marrow function:

     Absolute count of neutrophil ≥1.5×10^9/L; Platelet count ≥90×10^9/L; Hemoglobin ≥ 90g/L; AST, ALT≤2.5×ULN (subjects with liver metastasis ≤5×ULN); Totol bilirubin ≤1.5×ULN（Gilbert syndrome≤3×ULN）; Serum creatinine ≤1.5×ULN, or estimated creatinine clearance (CrCl)≥60 mL/min (Cockcroft-Gault formula); Activated partial thromboplastin time (APTT) ≤1.5×ULN, while international normalized ratio (INR) or prothrombin (PT) ≤1.5×ULN;
  8. Left ventricular ejection fraction (LVEF) ≥ 50% detected by echocardiography; Arrhythmias that do not require treatment, the QT interval (QTcF) corrected by the Fridericia method is ≤ 470 ms (QTcF is calculated using the Fridericia formula, i.e. QTcF=QT/(RR ^ 0.33), RR is the standardized heart rate value, RR=60/heart rate); If there is an abnormality during the first inspection, it can be retested twice with an interval of at least 5 minutes, and the overall result/average value should be taken to determine the qualification; Basic blood oxygen saturation in indoor natural air environment>91%;
  9. Test subjects must have recovered from all prior therapy-related toxicities to ≤Grade 1 according to Common Terminology Criteria for Adverse Events (CTCAE) v5.0; except for alopecia (tumor resection);
  10. Test subjects with child-bearing potential must be willing to practice approved highly effective methods of contraception at the time of informed consent, and continue within 1 year after the completion of treatment;
  11. Be able to understand and sign the informed consent document.

Exclusion Criteria:

* Patients with any of the following criteria will not be allowed to participation:

  1. Test subjects who have a history of hypersensitivity to any component or excipient of HS-IT101 or other study drugs (cyclophosphamide, fludarabine and recombinant human interleukin-2);
  2. Test subjects have any uncontrollable clinical problems (including but not limited):

     hypertension poorly controlled by medication (blood pressure ≥160/100mmHg at rest after taking medication); poorly controlled diabetes; cardiac disease (New York Heart Association class Ⅲ/Ⅳ congestive heart failure or heart block);
  3. Test subjects who have active major medical illnesse(es) of the cardiovascular (within 6 months prior to enrollment), including deep vein thrombosis or pulmonary embolism; myocardial infarction; severe or unstable arrhythmia or angina pectoris; percutaneous coronary intervention, acute coronary syndrome, coronary artery bypass grafting; cerebrovascular accident, transient cerebral ischemia Seizures, cerebral embolism;
  4. Active autoimmune diseases that require systemic treatment during the study period (eczema, vitiligo, psoriasis, alopecia or Grave's disease that do not require systematic treatment in the past two years, other autoimmune diseases that are not expected to recur, hypothyroidism that only requires thyroid hormone replacement therapy, and type I diabetes subjects that only require insulin replacement therapy can be included);
  5. Organ transplantation and a history of hematopoietic stem cell transplantation;
  6. Any immunosuppressive drugs, such as steroids, have been used within 4 weeks prior to tumor tissue sampling, or the researcher has determined the presence of comorbidities that require the use of immunosuppressive drugs during the trial period. However, physiological doses of glucocorticoids (i.e. ≤ 12 mg/m2/day of hydrocortisone or other hormones within the equivalent dose range after equivalent dose conversion) are allowed, and steroid drugs are allowed for intranasal or local use;
  7. Individuals who have received systematic anti-tumor therapy within 4 weeks prior to pre-treatment (including those who have participated in other clinical trial drug treatments; those who have metabolized 5 drugs with a half-life of less than 4 weeks, whichever is shorter) or those who plan to participate in other intervention clinical trials during the study period;
  8. Presence of acute or chronic infection:

     HIV positive, Treponema pallidum antibody positive, or clinically active hepatitis B and C, including virus carriers (excluding HBsAg and/or HBeAg positive individuals for hepatitis B; excluding HCVAb positive individuals for hepatitis C);Active infections or active tuberculosis infections that require systemic treatment;
  9. Vaccinated with the new coronavirus vaccine within 4 weeks propr to screening, or who have received a live vaccine within 3 months, or who plan to receive live vaccine during the trial;
  10. Major organs underwent surgery (excluding needle biopsy) or significant trauma within 4 weeks before screening；required elective surgery during the study;
  11. Patients who have surgical complications or delayed healing prior to screening, and have been determined by the researchers to increase the risk of gonorrhea pretreatment, adoptive TIL therapy, and IL-2 adjuvant therapy;
  12. Test subjects who have had another primary malignancy within the previous 5 years, excluding basal cell carcinoma of the skin, squamous cell carcinoma of the skin and/or carcinoma in situ after radical resection;
  13. Suffering from severe respiratory system diseases (with a history of or combined with severe interstitial lung disease, severe chronic obstructive pulmonary disease, severe pulmonary insufficiency, and symptomatic bronchospasm);
  14. Patients with gastrointestinal bleeding requiring surgical treatment, local intestinal ischemia or perforation;
  15. Patients with known meninges metastasis; Patients with known uncontrolled or untreated central nervous system metastases (excluding those who have received stable treatment symptoms and stopped glucocorticoid and anticonvulsant drug treatment ≥ 4 weeks prior to pre-treatment);
  16. Previously received similar cell therapy products;
  17. Females in pregnancy or lactation;
  18. Subject have mental illness, alcoholism, drug or substance abuse；or researchers considering the test subject as having other reasons inappropriate for the clinical study.

Ages: 18 Days to 75 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 44 (Estimated)
Dates: Start 2024-01-18 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2028-03-31 (Estimated)

PRIMARY OUTCOMES:
Adverse Events (AE) | 12 months
  To characterize the safety profile of HS-IT101 in patients with advanced solid tumor as assessed by incidence of adverse events
Serious Adverse Events (SAE) | 12 months
  To characterize the safety profile of HS-IT101 in patients with advanced solid tumor as assessed by incidence of serious adverse events

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | Up to 36 months
  To evaluate the efficacy of HS-IT101 in patients with advanced solid tumor, based on the objective response rate (ORR) as assessed by the Independent Review Committee (IRC) per RECIST v1.1
Time-to-response (TTR) | Up to 36 months
  To evaluate the efficacy of HS-IT101 in patients with advanced solid tumor by assessing the time-to-response (TTR) as assessed by the Investigator per RECIST v1.1
Duration of Response (DOR) | Up to 36 months
  To evaluate the efficacy of HS-IT101 in patients with advanced solid tumor by assessing the duration of response (DOR) as assessed by the Investigator per RECIST v1.1
Disease Control Rate (DCR) | Up to 36 months
  To evaluate the efficacy of HS-IT101 in patients with advanced solid tumor, based on the disease control rate (DCR) as assessed by the Independent Review Committee (IRC) per RECIST v1.1
Progression-Free-Survival (PFS) | Up to 36 months
  To evaluate progression-free-survival (PFS) in patients with advanced solid tumor
Overall Survival (OS) | Up to 36 months
  To evaluate overall survival (OS) in patients with advanced solid tumor
Lymphocyte subpopulation | Up to 6 months
  Percentage and absolute count of T, B,NK cells
TCR repertoire | Up to 6 months
  VDJ recombination of the different TCR genes

CONTACTS AND LOCATIONS:
Overall Officials: Ning Li, MD, Principal Investigator — Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Locations (1):
- Cancer Hospital, Chinese Academy of Medical Sciences, Beijing, Beijing Municipality, China